CLINICAL TRIAL: NCT06165003
Title: Examining the Effect of Nurses' Use of Broselow Tape in Non-resuscitation Pediatric Emergency Department Practices on Patient Safety
Brief Title: Examination of Nurses' Use of Broselow Tape in Non-resuscitation Pediatric Emergency Department Practices
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Aslı Alaca, Principal İnvestigator, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Aslı alaca
Record Dates: First submitted 2023-11-25; First posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Pediatric
Keywords: broselow tape; pediatric emergency department; nurse

STUDY DESIGN:
Intervention Model Description: Randomized controlled study
Who Masked: Participant
Masking Description: In the research, control group data will be collected first. After the data of the control group is collected, the data of the experimental group will be collected.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Peripheral Intravenous Catheter Insertion Procedure - Broselow Band Selection - Experimental Group Urinary Catheter Insertion Procedure - Broselow Tape Selection - Experimental Group Aspiration process - Broselow Band Selection - Experimental group Nasogastric/Orogastric Catheter Insertion Procedure - Broselow Band Selection - Experimental Group
  Interventions: Other: Use of broselow tape
- Control Group (No Intervention): Peripheral Intravenous Catheter Insertion Procedure - Routine Application - Control Group Urinary Catheter Insertion Procedure - Routine Application - Control Group Aspiration process - Routine Application - Control Group Nasogastric/Orogastric Catheter Insertion Procedure - Routine Practice - Control Group

INTERVENTIONS:
Other: Use of broselow tape — In the research, the nurse is the decision maker in the selection of the catheters to be used in the procedures (peripheral intravenous catheter insertion, urinary catheter insertion, aspiration procedure, nasogastric/orogastric catheter insertion) for the patients in the control group.
  In these procedures, the nurse's choices will be evaluated as control group data as routine clinical practice.
  After the control group data is collected, Broselow tape will be used in the selection of catheters to be used in the procedures to be performed on the patients in the experimental group (peripheral intravenous catheter insertion, urinary catheter insertion, aspiration procedure, nasogastric/orogastric catheter insertion).
  Our research will be conducted to examine the effect of nurses' use of Broselow tape in non-resuscitation applications and to minimize errors and application disruptions in procedures involving nurses.
  Arms: Experimental group

SUMMARY:
The patient's body weight is often taken as a basis when calculating drug doses and determining equipment sizes for pediatric patients presenting to the emergency department.

The methods used to determine body weight are the family's estimated weight, formulas for estimating weight according to age, or the Broselow band used to estimate weight according to height.

Weight estimates that are incomplete compared to the child's actual body weight lead to medication errors, wrong material selection and prolongation of the procedure, resulting in increased mortality and morbidity.

DETAILED DESCRIPTION:
This study will be carried out to create an evidence-based practice in the selection of catheters to be used during peripheral intravenous catheter insertion, urinary catheter insertion, nasogastric/orogastric catheter insertion and aspiration in children using the Broselow band in non-resuscitation applications coming to the Pediatric Emergency Department.

By using the Boselow band in non-resuscitation pediatric emergency department applications, reducing the number of attempts and errors by ensuring the correct equipment selection in the procedures applied to patients, and increasing the success of the procedure; This will be done to ensure that the decisions taken by nurses using their experience and previous knowledge are more systematic.

ELIGIBILITY:
Inclusion Criteria:

* Children weighing 3 to 36 kg and 47 to 143 cm tall
* Children aged 0-18
* Patients coming to the emergency department for non-resuscitation procedures
* Patients and their families who volunteer to participate in the research
* Patients who will have a peripheral intravenous catheter inserted
* Patients who will have a urinary catheter inserted
* Patients who will have a nasogastric/orogastric catheter inserted
* Patients who will undergo aspiration procedure

Exclusion Criteria:

* Children weighing less than 3 kg and taller than 143 cm
* Children with anomaly contractures that may prevent measurement during measurement with the Broselow tape
* Patients with central venous catheter
* Patients with peripheral intravenous catheters outside the pediatric emergency department
* Patients who have a urinary catheter inserted outside the pediatric emergency department
* Patients who have a nasogastric/orogastric catheter inserted outside the pediatric emergency department

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 246 (Estimated)
Dates: Start 2023-11-30 (Estimated); Primary Completion 2024-06-26 (Estimated); Study Completion 2025-12-26 (Estimated)

PRIMARY OUTCOMES:
Selection by broselow Band | 2 year
  Success of Broselow band selection

SECONDARY OUTCOMES:
Nurses' success rate in catheter applications | 2 year
  Number of attempts
Nurses' success rate in catheter applications | 2 year
  length of stay of the catheters
Nurses' success rate in catheter applications | 2 year
  nurses' completion of the catheter insertion process

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Argall JA, Wright N, Mackway-Jones K, Jackson R. A comparison of two commonly used methods of weight estimation. Arch Dis Child. 2003 Sep;88(9):789-90. doi: 10.1136/adc.88.9.789. No abstract available. PMID 12937099
- [Background] Luscombe M, Owens B. Weight estimation in resuscitation: is the current formula still valid? Arch Dis Child. 2007 May;92(5):412-5. doi: 10.1136/adc.2006.107284. Epub 2007 Jan 9. PMID 17213259
- [Derived] Alaca A, Sari HY. An examination of how nurses' use of the Broselow tape affects patient safety during peripheral intravenous catheterization. Int Emerg Nurs. 2026 Feb;84:101712. doi: 10.1016/j.ienj.2025.101712. Epub 2025 Nov 25. PMID 41297189